CLINICAL TRIAL: NCT00112957
Title: Phase II Study of Recombinant Vaccinia-NY-ESO-1 (rV-NY-ESO-1) and Recombinant Fowlpox-NY-ESO-1 (rF-NY-ESO-1) in Patients With Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma Whose Tumors Express NY-ESO-1 or LAGE-1 Antigen
Brief Title: Vaccine Therapy in Patients With Stage II, III, or IV Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD 2002-012; RPCI-I-13303; CDR0000424461
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: fallopian tube cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- rV- and rF-NY-ESO-1 (Experimental): Patients received a single intradermal injection of rV-NY-ESO-1 (3.1 × 10^7 PFU) on Day 1, followed by subcutaneous injections of rF-NY-ESO-1 (7.41 × 10^7 PFU) on Days 29, 57, 85, 113, 141, and 169 or until observation of treatment-related ≥ grade 3 toxicity or disease progression.
  Interventions: Biological: rV-NY-ESO-1 vaccine; Biological: rF-NY-ESO-1 vaccine

INTERVENTIONS:
Biological: rV-NY-ESO-1 vaccine — Patients received a single intradermal injection of rV-NY-ESO-1 (3.1 × 10^7 PFU) on Day 1.
Biological: rF-NY-ESO-1 vaccine — Patients received subcutaneous injections of rF-NY-ESO-1 (7.41 × 10^7 PFU) on Days 29, 57, 85, 113, 141, and 169.

SUMMARY:
This was a Phase 2, single-center, open-label study of recombinant vaccinia-NY-ESO-1 (rV-NY-ESO-1) and recombinant fowlpox-NY-ESO-1 (rF-NY-ESO-1) injections in patients who had a complete response to standard therapy for epithelial ovarian, fallopian tube, or primary peritoneal carcinoma and whose tumors expressed NY-ESO-1 or LAGE-1 antigen. Study objectives were to evaluate maintenance of remission at 12 months, time to failure of vaccine therapy, cellular and humoral immunity and any correlation with time to failure, and safety.

DETAILED DESCRIPTION:
Patients received a single intradermal injection of rV-NY-ESO-1 (3.1 × 10^7 plaque forming units [PFU]) on Day 1, followed by monthly subcutaneous injections of rF-NY-ESO-1 (7.41 × 10^7 PFU) for 6 months (Days 29, 57, 85, 113, 141, and 169) or until observation of treatment-related ≥ grade 3 toxicity or disease progression. Study injections were administered during a 28-week evaluation period. Patients returned to the clinic for follow-up on Day 197 (i.e., 28 days after the last study injection) and every 2 months thereafter for at least 12 months. In patients with measurable disease, tumor response was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. Patients were monitored continuously for safety for the duration of study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented epithelial carcinoma arising in the ovary, fallopian tube, or peritoneum, from stage II to IV at diagnosis.
2. Received initial surgery and chemotherapy with at least one platinum-based chemotherapy regimen.
3. Demonstrated complete response to first line therapy as evidenced by negative clinical examination, cancer antigen (CA)-125 tumor marker, and computed tomography (CT) scan. In addition, if second-look surgery was performed, patients must have had no evidence of microscopic or macroscopic disease. Patients must have been within 6 months of completing their first line platinum-based chemotherapy. These patients would normally enter a period of observation as standard management.
4. Tumor expression of 1) NY-ESO-1 by reverse transcription-polymerase chain reaction (RT-PCR) analysis, preferably, or immunohistochemistry; or 2) LAGE-1 by RT-PCR.
5. Expected survival of at least 6 months.
6. Full recovery from surgery.
7. Karnofsky performance status of 70% or more.
8. Patients must have had the following clinical laboratory results:

   * neutrophil count: ≥ 1.5 x 10^9/L
   * lymphocyte count: ≥ 0.5 x 10^9/L
   * platelet count: ≥ 100 x 10^9/L
   * serum creatinine: ≤ 2 mg/dL
   * serum bilirubin: ≤ 2 mg/dL
9. Ability to avoid close contact with children < 3 years of age; pregnant or breast feeding women; individuals with active, or a history of, eczema or atopic dermatitis or other skin disorders such as burns, chickenpox, shingles, impetigo, herpes, severe acne, or psoriasis; and immunocompromised individuals (human immunodeficiency virus [HIV], leukemia, lymphoma, solid organ transplantation, generalized malignancy, cellular or humoral immunodeficiency syndromes, patients currently receiving cytotoxic chemotherapies, radiation, or high dose corticosteroids).
10. Have been informed of other treatment options.
11. Age ≥ 18 years.
12. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may have been available.
2. Other serious illnesses (eg, serious infections requiring antibiotics, bleeding disorders).
3. History of current eczema or atopic dermatitis.
4. History of autoimmune disease (eg., thyroiditis, lupus).
5. Other acute, chronic, or exfoliative skin conditions such as burns, chickenpox, shingles, impetigo, herpes, severe acne, or psoriasis.
6. Concomitant systemic treatment with corticosteroids, anti-histamine or non-steroidal anti-inflammatory drugs. Specific cyclooxygenase-2 inhibitors were permitted.
7. Chemotherapy, radiation therapy, or immunotherapy within 4 weeks before study entry (6 weeks for nitrosoureas).
8. Known HIV positivity.
9. Known allergy or severe reaction to a smallpox (vaccinia) vaccination.
10. Known allergy to eggs, determined by history.
11. Myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, chest pain or shortness of breath with activity, or other heart conditions being treated by a doctor.
12. Presence of 3 or more of the following risk factors:

    * Hypertension
    * Hypercholesterolemia
    * Diabetes
    * A first degree relative (for example, mother, father, brother, sister) who had a heart condition before the age of 50
    * Current cigarette smoker
13. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
14. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
15. Lack of availability of a patient for immunological and clinical follow-up assessment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rV- and rF-NY-ESO-1
Started | 23
Completed (Completed through the 12-month follow-up) | 4
Not Completed | 19
Not completed — Progressive disease | 18
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set includes all patients who received at least 1 injection with rV-NY-ESO-1 or rF-NY-ESO-1.
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 55 [37 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
Karnofsky Performance Status [Count of Participants; unit: Participants] — Functional impairment is as follows: 100=normal, no complaints; 90=able to carry on normal activities with minor signs/symptoms of disease; 80=normal activity with effort; 70=care for self, unable to carry on normal activity or to do active work; 60=requires occasional assistance, but able to care for most needs; 50=requires considerable assistance & frequent medical care; 40=disabled, requires special care and assistance; 30=severly disabled, hospitalization indicated though death nonimminent; 20=very sick, hospitalization necessary, active supportive treatment necessary; 10=moribund; 0=dead
  Participants
    70 | 1
    80 | 3
    90 | 3
    100 | 16
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients in Remission at 1 Year
Description: Time to failure (TTF) was evaluated as the crude proportion of patients in remission at 1 year, calculated as: 100 x (number of patients in remission at 1 year)/(number of patients with known status at 1 year). The Kaplan-Meier cumulative estimate of the proportion of patients in remission at 1 year was also calculated.
Time Frame: 12 months
Population: The Full Analysis Set includes all patients who received at least 1 injection with rV-NY-ESO-1 or rF-NY-ESO-1 and met the entry criterion of having epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. One patient with breast cancer was treated in the protocol under compassionate use and is excluded from the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 22
percentage of participants
  Crude rate: number analyzed (Participants) | 21
  Crude rate | 38.1 [18.1 to 61.6]
  Kaplan-Meier cumulative rate: number analyzed (Participants) | 21
  Kaplan-Meier cumulative rate | 38.8 [18.8 to 58.5]

2. Secondary Outcome: Mean Time to Failure Among Patients Who Progressed On Study
Description: TTF was calculated as the number of days from the first dose until the patient discontinued due to progressive disease. Patients who completed the study or discontinued for other reasons were considered censored at the day of their last study visit, including the follow-up visits after Day 197. Progression was defined using the Response Evaluation Criteria In Solid Tumors (RECIST [version 1.0]) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 20 months
Population: The Full Analysis Set includes all patients who received at least 1 injection with rV-NY-ESO-1 or rF-NY-ESO-1 and met the entry criterion of having epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. TTF was calculated for the subset of patients who had disease progression at any time.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 17
days | 253.1 (160.4)

3. Secondary Outcome: Number of Patients With Best Overall Tumor Response
Description: Tumor responses were evaluated using computed tomography and were categorized according to RECIST (version 1.0) at Screening, on Days 85 and 197 and every 2 months thereafter for at least 12 months. Per RECIST, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions (no evaluable disease); Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 22
Participants
  Response at Day 85: Stable Disease | 3
  Response at Day 85: Progressive Disease | 0
  Response at Day 85: No Evaluable Disease | 15
  Response at Day 85: Missing/Not Done | 4
  Response at Day 197: Stable Disease | 3
  Response at Day 197: Progressive Disease | 1
  Response at Day 197: No Evaluable Disease | 11
  Response at Day 197: Missing/Not Done | 7
  Response at 12-Month Follow-up: Stable Disease | 0
  Response at 12-Month Follow-up: Progressive Disease | 0
  Response at 12-Month Follow-up: No Evaluable Disease | 4
  Response at 12-Month Follow-up: Missing/Not Done | 18
  Response at End of Study: Stable Disease | 3
  Response at End of Study: Progressive Disease | 4
  Response at End of Study: No Evaluable Disease | 0
  Response at End of Study: Missing/Not Done | 15

4. Secondary Outcome: Mean Absolute Cancer Antigen-125 Values Over Time on Study
Description: Blood samples were collected to measure serum levels of tumor marker cancer antigen (CA)-125 at Screening and on Days 1, 29, 57, 85, 113, 141, 169, and 197 and every 2 months for at least 12 months following Day 197.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 22
U/mL
  CA-125 at Baseline | 17.9 (15.4)
  CA-125 at Day 29 | 27.5 (40.7)
  CA-125 at Day 57: number analyzed (Participants) | 21
  CA-125 at Day 57 | 74.8 (203.7)
  CA-125 at Day 85: number analyzed (Participants) | 18
  CA-125 at Day 85 | 12.8 (9.6)
  CA-125 at Day 113: number analyzed (Participants) | 18
  CA-125 at Day 113 | 20.4 (33.6)
  CA-125 at Day 141: number analyzed (Participants) | 16
  CA-125 at Day 141 | 11.8 (7.2)
  CA-125 at Day 169: number analyzed (Participants) | 16
  CA-125 at Day 169 | 14.1 (9.3)
  CA-125 at Day 197: number analyzed (Participants) | 15
  CA-125 at Day 197 | 16.0 (13.4)
  Follow-up at Month 2: number analyzed (Participants) | 13
  Follow-up at Month 2 | 80.7 (205.9)
  Follow-up at Month 4: number analyzed (Participants) | 9
  Follow-up at Month 4 | 16.0 (14.6)
  Follow-up at Month 6: number analyzed (Participants) | 7
  Follow-up at Month 6 | 80.4 (187.2)
  Follow-up at Month 8: number analyzed (Participants) | 6
  Follow-up at Month 8 | 10.6 (3.5)
  Follow-up at Month 10: number analyzed (Participants) | 6
  Follow-up at Month 10 | 59.5 (120.5)
  Follow-up at Month 12: number analyzed (Participants) | 4
  Follow-up at Month 12 | 16.8 (12.6)

5. Secondary Outcome: Number of Patients With NY-ESO-1 and LAGE-1-specific Immunity
Description: Specific antibody response to the NY-ESO-1 and LAGE-1 antigen was measured by enzyme-linked immunosorbent assay (ELISA) at Screening, Days 29, 57, 85, 113, 141, 169, 197, Month 6, and Month 12.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 22
Participants
  Screening: NY-ESO-1 Positive | 3
  Screening: LAGE-1 Positive | 2
  Day 29: NY-ESO-1 Positive | 7
  Day 29: LAGE-1 Positive | 5
  Day 57: NY-ESO-1 Positive: number analyzed (Participants) | 21
  Day 57: NY-ESO-1 Positive | 6
  Day 57: LAGE-1 Positive: number analyzed (Participants) | 21
  Day 57: LAGE-1 Positive | 4
  Day 85: NY-ESO-1 Positive: number analyzed (Participants) | 18
  Day 85: NY-ESO-1 Positive | 5
  Day 85: LAGE-1 Positive: number analyzed (Participants) | 18
  Day 85: LAGE-1 Positive | 4
  Day 113: NY-ESO-1 Positive: number analyzed (Participants) | 18
  Day 113: NY-ESO-1 Positive | 6
  Day 113: LAGE-1 Positive: number analyzed (Participants) | 18
  Day 113: LAGE-1 Positive | 3
  Day 141: NY-ESO-1 Positive: number analyzed (Participants) | 16
  Day 141: NY-ESO-1 Positive | 5
  Day 141: LAGE-1 Positive: number analyzed (Participants) | 16
  Day 141: LAGE-1 Positive | 3
  Day 169: NY-ESO-1 Positive: number analyzed (Participants) | 16
  Day 169: NY-ESO-1 Positive | 5
  Day 169: LAGE-1 Positive: number analyzed (Participants) | 16
  Day 169: LAGE-1 Positive | 3
  Day 197: NY-ESO-1 Positive: number analyzed (Participants) | 15
  Day 197: NY-ESO-1 Positive | 5
  Day 197: LAGE-1 Positive: number analyzed (Participants) | 15
  Day 197: LAGE-1 Positive | 3
  Month 6: NY-ESO-1 Positive: number analyzed (Participants) | 8
  Month 6: NY-ESO-1 Positive | 4
  Month 6: LAGE-1 Positive: number analyzed (Participants) | 8
  Month 6: LAGE-1 Positive | 0
  Month 12: NY-ESO-1 Positive: number analyzed (Participants) | 4
  Month 12: NY-ESO-1 Positive | 1
  Month 12: LAGE-1 Positive: number analyzed (Participants) | 4
  Month 12: LAGE-1 Positive | 1

6. Secondary Outcome: Number of Patients With Release of Interferon-Gamma by T Cells in Response to Cancer Antigens
Description: Intracellular cytokine staining assays were performed at Screening, Days 85 and 197, Month 6, and Month 12 to evaluate the release of interferon-gamma by CD4 and CD8 T cells following study injections.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 22
Participants
  Screening: CD4: Positive | 10
  Screening: CD4: Negative | 12
  Screening: CD8: Positive | 2
  Screening: CD8: Negative | 20
  Day 85: CD4: number analyzed (Participants) | 18
  Day 85: CD4: Positive | 13
  Day 85: CD4: Negative | 5
  Day 85: CD8: number analyzed (Participants) | 18
  Day 85: CD8: Positive | 6
  Day 85: CD8: Negative | 12
  Day 197: CD4: number analyzed (Participants) | 15
  Day 197: CD4: Positive | 12
  Day 197: CD4: Negative | 3
  Day 197: CD8: number analyzed (Participants) | 14
  Day 197: CD8: Positive | 5
  Day 197: CD8: Negative | 9
  Month 6: CD4: number analyzed (Participants) | 8
  Month 6: CD4: Positive | 6
  Month 6: CD4: Negative | 2
  Month 6: CD8: number analyzed (Participants) | 8
  Month 6: CD8: Positive | 3
  Month 6: CD8: Negative | 5
  Month 12: CD4: number analyzed (Participants) | 4
  Month 12: CD4: Positive | 3
  Month 12: CD4: Negative | 1
  Month 12: CD8: number analyzed (Participants) | 4
  Month 12: CD8: Positive | 1
  Month 12: CD8: Negative | 3

7. Secondary Outcome: Number of Patients With Detectable T-cell Responses Following Vaccination
Description: NY-ESO-1-specific CD8+ T cells (human leukocyte antigen [HLA]-A2 patients only) and NY-ESO-1-specific CD4+ T cells (HLA-DP4 patients only) were measured by interferon-gamma enzyme-linked immunosorbent spot (ELISPOT) assay. The response to the ELISPOT assay was considered to be positive if the number of spots in the peptide-exposed well was 2-fold or more higher than the number of spots in the unstimulated well, and if there was a minimum of 10 (after subtraction of background spots) peptide-specific spots/25,000 T-cells, or less if T-cell clones were used.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 22
Participants
  Detectable CD4+ T-cell response | 20
  Detectable CD8+ T-cell response | 10

8. Secondary Outcome: Number of Patients With Delayed-Type Hypersensitivity Reactions Following Vaccination
Description: NY-ESO-1 antigen-specific delayed-type hypersensitivity (DTH) was measured by skin test at Screening and on Days 113 and 197. All patients were tested for the NY-ESO-1 protein, with additional DTH testing as follows: patients who were HLA-A2+ had NY-ESO-1b testing, patients who were HLA-DP4+ had NY-ESO-DP4 testing, and patients who were both HLA-A2+ and HLA-DP4+ had NY-ESO-1b and NY-ESO-DP4 testing.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 22
Participants
  NY-ESO-1 protein: Induration at Screening | 1
  NY-ESO-1 protein: Redness at Screening | 5
  NY-ESO-1 protein: Induration at Day 113: number analyzed (Participants) | 18
  NY-ESO-1 protein: Induration at Day 113 | 1
  NY-ESO-1 protein: Redness at Day 113: number analyzed (Participants) | 18
  NY-ESO-1 protein: Redness at Day 113 | 4
  NY-ESO-1 protein: Induration at Day 197: number analyzed (Participants) | 15
  NY-ESO-1 protein: Induration at Day 197 | 0
  NY-ESO-1 protein: Redness at Day 197: number analyzed (Participants) | 15
  NY-ESO-1 protein: Redness at Day 197 | 1
  NY-ESO-1b: Induration at Screening | 1
  NY-ESO-1b: Redness at Screening | 1
  NY-ESO-1b: Induration at Day 113: number analyzed (Participants) | 18
  NY-ESO-1b: Induration at Day 113 | 0
  NY-ESO-1b: Redness at Day 113: number analyzed (Participants) | 18
  NY-ESO-1b: Redness at Day 113 | 0
  NY-ESO-1b: Induration at Day 197: number analyzed (Participants) | 15
  NY-ESO-1b: Induration at Day 197 | 0
  NY-ESO-1b: Redness at Day 197: number analyzed (Participants) | 15
  NY-ESO-1b: Redness at Day 197 | 0
  NY-ESO-DP4: Induration at Screening | 0
  NY-ESO-DP4: Redness at Screening | 2
  NY-ESO-DP4: Induration at Day 113: number analyzed (Participants) | 18
  NY-ESO-DP4: Induration at Day 113 | 0
  NY-ESO-DP4: Redness at Day 113: number analyzed (Participants) | 18
  NY-ESO-DP4: Redness at Day 113 | 0
  NY-ESO-DP4: Induration at Day 197: number analyzed (Participants) | 15
  NY-ESO-DP4: Induration at Day 197 | 0
  NY-ESO-DP4: Redness at Day 197: number analyzed (Participants) | 15
  NY-ESO-DP4: Redness at Day 197 | 0

9. Secondary Outcome: Number of Patients With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), version 3.0. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the study period.
Time Frame: Continuously for up to 20 months
Population: The Safety Analysis Set includes all patients who received at least 1 injection with rV-NY-ESO-1 or rF-NY-ESO-1.
Measure: Count of Participants; unit: Participants
Arm/Group | rV- and rF-NY-ESO-1
Number analyzed (Participants) | 23
Participants
  Any TEAE | 23
  Maximum grade 1 TEAE | 3
  Maximum grade 2 TEAE | 15
  Maximum grade 3 TEAE | 3
  Maximum grade 4 TEAE | 2
  Treatment-related TEAE | 9
  Serious TEAE | 4
  TEAE Leading to Treatment Discontinuation | 2

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 20 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTC (version 3.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per patient at the maximum reported grade.
Arm/Group | rV- and rF-NY-ESO-1
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 4/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rV- and rF-NY-ESO-1 (N=23)
Urinary tract infection (Infections and infestations) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Pneumonia (Infections and infestations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Septic shock (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rV- and rF-NY-ESO-1 (N=23)
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 3
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 2
Injection site pruritus (General disorders) | 2
Injection site reaction (General disorders) | 2
Injection site scab (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Skin test positive (Investigations) | 20
Blood creatinine increased (Investigations) | 2
Blood glucose increased (Investigations) | 2
Blood urea increased (Investigations) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 3
Pollakiuria (Renal and urinary disorders) | 2
Breast tenderness (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less